CLINICAL TRIAL: NCT00309127
Title: A Multicentre, Randomised Study to Examine the Effects of Disease Management on Development of End Stage Renal Disease in Type 2 Diabetic Patients With Nephropathy
Brief Title: Effects of Disease Management on Development of End Stage Renal Disease in Type 2 Diabetic Patients With Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Juliana Chan, Chair Professor of Medicine and Therapeutics, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2004.226-T; HCPF No. 121012
Record Dates: First submitted 2006-03-30; First posted 2006-03-31 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Type 2 Diabetes Mellitus; DM Nephropathy
Keywords: Type 2 Diabetes Mellitus; DM Nephropathy; Structured care
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Patient Care Team

INTERVENTIONS:
Behavioral: Multidisciplinary team care

SUMMARY:
Disease management using a multidisciplinary team to achieve and maintain optimal metabolic and cardiovascular risk factors control in Type 2 diabetic patients with nephropathy reduces the incidence of end stage renal disease (ESRD) and improves clinical outcomes compared to usual clinic-based care

DETAILED DESCRIPTION:
Diabetic patients consume over 10% of health care costs in most developed countries. Over 80% of these resources are used to treat diabetic complications and late stage diseases. Over 30% of patients admitted to the medical wards in Hong Kong's public hospitals have diabetes, mainly due to cardiovascular and renal complications. Diabetes is now the leading cause of end stage renal disease (ESRD), accounting for 30-50% of patients on renal replacement therapy (RRT). In Hong Kong, the number of patients receiving RRT have increased by 50% in the last 5 years but the number of patients with ESRD due to diabetes have doubled. Between 10% and 15% of patients attending medical clinics in local public hospitals either receive insulin or anti-diabetic drugs. In both community and hospital settings, between 30% and 50% of diabetic patients have albuminuria, which is by far the most powerful predictor for early mortality, cardiovascular morbidity and renal disease. Local published data show that 3-10% of diabetic patients died or developed clinical endpoints yearly.

There are now overwhelming evidence supporting the beneficial effects of optimal control of cardiovascular risk factors on clinical outcomes in diabetic patients. However, there are few studies to examine the most effective way to translate these scientific evidence collected in closely monitored clinical trial situations into daily clinical practice. Results from this multi-centre, randomized study will provide important information to health care policy makers regarding the cost effectiveness of disease management using a multidisciplinary team to deliver a structured care model in light of the growing diabetes epidemic and the constraints of finite resources and the need for equity.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetic patients with ages between 35 and 75 years (inclusive) and defined according to the 1998 WHO criteria and no history of unprovoked ketosis and not requiring continuous insulin treatment within 1 year of diagnosis
2. Plasma creatinine 150-350 mmol/l (inclusive) who had no microscopic haematuria and no ultrasonographic evidence of obstructive uropathy which is amenable to surgical intervention

Exclusion Criteria:

1. patients with malignancy or other life-threatening diseases
2. ultrasonographic evidence of obstructive uropathy which is amenable to surgical intervention
3. non-diabetes related renal disease such as glomerulonephritis proven on renal biopsy reversible kidney disease, to be ruled out by ultrasonographic examination
4. patients with clinically unstable psychiatric illnesses
5. Patients who have 2 consecutive values of plasma creatinine concentration which differ by more than 20% within 3 months prior to recruitment.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2003-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Death and/or ESRD defined as need for dialysis or plasma creatinine 500mmol/l | May 2003 - Dec 2007

SECONDARY OUTCOMES:
Composite cardiovascular endpoints (acute myocardial infarction, revascularisation procedures, heart failure or unstable angina or arrhythmia requiring hospital admissions, lower extremity amputation) | May 2003 - Dec 2007
Number of hospital admissions, total number of days of hospital stay and attendance at the Accident and Emergency Department | May 2003 - Dec 2007

CONTACTS AND LOCATIONS:
Overall Officials: Juliana CN Chan, MB ChB, MD, Principal Investigator — Department of Medicine and Therapeutics, The Chinese University of Hong Kong, The Prince of Wales Hospital, Shatin
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Cashmore BA, Cooper TE, Evangelidis NM, Green SC, Lopez-Vargas P, Tunnicliffe DJ. Education programmes for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 Aug 22;8(8):CD007374. doi: 10.1002/14651858.CD007374.pub3. PMID 39171639
- [Derived] Chan JC, So WY, Yeung CY, Ko GT, Lau IT, Tsang MW, Lau KP, Siu SC, Li JK, Yeung VT, Leung WY, Tong PC; SURE Study Group. Effects of structured versus usual care on renal endpoint in type 2 diabetes: the SURE study: a randomized multicenter translational study. Diabetes Care. 2009 Jun;32(6):977-82. doi: 10.2337/dc08-1908. PMID 19460913